CLINICAL TRIAL: NCT01846182
Title: RCT of Duloxetine & Pregabalin for the Treatment of Gulf War Illness in Veterans
Brief Title: Research Examining Gulf War Illness in Our Nations Service Members
Acronym: REGIONS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated by Funder
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPLD-016-12F; 6125 (Other: Clinical Science Research & Development)
Record Dates: First submitted 2013-04-16; First posted 2013-05-03 (Estimated); Results first posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-02

CONDITIONS: Gulf War Illness
Keywords: Gulf War Illness; Pregabalin; Duloxetine; Gulf War Veterans; Cymbalta; Lyrica
MeSH Terms: interventions — Duloxetine Hydrochloride; Pregabalin

STUDY DESIGN:
Intervention Model Description: Three arms comparing placebo to duloxetine and pregabalin
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Active Comparator): 60 mg of duloxetine in the AM for 20 weeks and placebo in PM
  Interventions: Drug: Duloxetine; Drug: Placebo
- Group 2 (Active Comparator): 300 mg of pregabalin in the PM for 20 weeks and placebo in AM
  Interventions: Drug: Pregabalin; Drug: Placebo
- Group 3 (Placebo Comparator): placebo in the AM & PM for 20 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — serotonin norepinephrine reuptake inhibitor
  Other Names: Cymbalta
  Arms: Group 1
Drug: Pregabalin — alpha-2-alpha subunit calcium channel ligand
  Other Names: Lyrica
  Arms: Group 2
Drug: Placebo — Placebo

SUMMARY:
At least 1 in 4 of the 700,000 U.S. Veterans who served in the 1990-1991 Gulf War suffer from Gulf War Illness (GWI). Despite considerable research, effective treatments remain elusive. GWI refers to a complex of symptoms that typically include widespread chronic pain, persistent headache, memory and concentration problems, gastrointestinal difficulties, sleep disturbances and unexplained fatigue. These symptoms are similar to that of fibromyalgia syndrome (FMS), another multi-symptom condition. Whereas, effective treatments for GWI have yet to be found, the FDA has approved duloxetine and pregabalin for the treatment of FMS. The lack of progress in finding effective treatments for GWI, and the similarities between GWI and FMS, provides a rationale for determining if these medications can provide relief to Veterans who suffer from GWI. This randomized controlled trial will test the efficacy of Duloxetine and Pregabalin for treating Gulf War Veterans who suffer from GWI.

DETAILED DESCRIPTION:
At least 1 in 4 of the 700,000 U.S. Veterans who served in the 1990-1991 Gulf War suffer from Gulf War Illness (GWI). Despite considerable research, effective treatments remain elusive. GWI refers to a complex of symptoms that typically include widespread chronic pain, persistent headache, memory and concentration problems, gastrointestinal difficulties, sleep disturbances and unexplained fatigue. This symptom profile is similar to that of fibromyalgia syndrome (FMS), a multi-symptom condition similar to GWI. Whereas, effective treatments for GWI have yet to be found, progress has been made in identifying medications to treat FMS. For example, the FDA has approved a number of medications including Duloxetine and Pregabalin for the treatment of FMS. Compared to placebo (PBO) Duloxetine (a serotonin norepinephrine reuptake inhibitor) and Pregabalin (an alpha-2-alpha-subunit calcium-channel ligand) significantly improved pain responses and fatigue. The capacity of Duloxetine to increase central levels of serotonin and norepinephrine as well as the more complex alterations of neurotransmitters and central nervous system (CNS) mediators of pain attributed to pregabalin are thought to be responsible for the medication's effects on pain, mood and sleep. Clinical practice and one open-label trial support the use of these medications in combination to achieve optimal symptom improvement amongst GWI sufferers; however, such combinations have not been formally tested in randomized controlled trials. The lack of progress in finding effective treatments for GWI, and the similarities between GWI and FMS, provides a rationale for determining if these FDA approved medications can provide significant symptomatic relief to Veterans who suffer from GWI. Central Texas is home to one of the highest number of Gulf War Veterans in the nation, thus the investigators' research team is ideally situated to conduct the proposed study. In a randomized, double-blind, controlled trial, 180 Veterans who meet defining criteria for GWI and whose symptom profile includes chronic widespread pain and sleep disturbances will be treated with one of the following medications; 1) AM Duloxetine+ PM placebo (PBO); 2) PM Pregabalin + AM PBO or 3) AM PBO + PM PBO. All active treatments will titrate from a lower dose in 2-week increments to the full therapeutic doses (FDA-approved for FMS). The outcome of the PBO double-dummy period will be compared statistically with 18 weeks of active therapy (weeks 5-22).

ELIGIBILITY:
Inclusion Criteria:

* Living in Central Texas near Killeen, Austin, Temple or Waco
* Served on active military duty and deployed to the Persian Gulf region for some period between August 1990 & July 1991
* English speaking and able to understand the consent form and study questionnaires
* Willing to be randomized to treatment and participate in 1-month follow up
* men & women between the ages of 43 to 70
* meet Kansas GWI case definition for the diagnosis of GWI
* report a baseline score > 4 on a 10-point Pain Visual Analog Scale (VAS)
* female participants of childbearing potential must test negative for pregnancy at the time of enrollment based on a urine pregnancy test and agree to use a reliable method of birth control (for example, oral contraceptives or Norplant; a reliable barrier method of birth control [diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam); intrauterine devices; partner with vasectomy; or abstinence) during the study and for 2 months following the last dose of the study drug. [Note that this inclusion criterion applies only to females of childbearing potential. Females of childbearing potential are defined as women not surgically sterilized and between menarche and 2 years post-menopause.]

Exclusion Criteria:

* Unstable or poorly controlled chronic medical illness such as Diabetes type-II, Hypertension (HTN), heart disease, endocrine disorders, narrow angle glaucoma
* Significant Central Nervous System disease including transient ischemic attacks (TIAs) or stroke, Dementia, syncopal episodes, severe head trauma, multiple sclerosis
* Serious or advanced heart disease or clinically relevant abnormal electrocardiogram (ECG), postural hypotension
* Untreated sleep apnea or body mass index placing patients at risk for undiagnosed sleep apnea (BMI> 35 kg/m2)
* Diabetes type-I and patients with Diabetes type-II associated with peripheral neuropathy, hepatitis, liver failure/cirrhosis
* End stage renal disease
* History of hypersensitivity reaction to pregabalin, duloxetine, venlafaxine; active treatment with duloxetine or pregabalin; History of failure of duloxetine or pregabalin at therapeutic doses; history of angioedema reaction to pregabalin
* Active systemic infectious disease such as tuberculosis and HIV, shingles
* Autoimmune mediated illnesses such as systemic lupus erythematosis, rheumatoid arthritis, scleroderma
* History of mental illness requiring hospitalization (depression, bipolar illness, post traumatic stress disorder, history of suicide attempts, psychosis, schizophrenia spectrum); Current major depression of dysthymia; patients lacking capacity to make medical decisions
* Use of monoamine oxidase inhibitors (MAOIs) within 2 weeks of evaluation; Active ongoing use of the following agents: desvenlafaxine, fenfluramine, linezolid, milnacipran, phentermine, tryptophan, tramadol, opiates
* Current (meets criterion within the last 6 months) for drug or alcohol dependence (except for nicotine and caffeine)
* Cancer other than non-melanoma skin cancers
* Women who are pregnant or desire to become pregnant, breastfeeding, who use unreliable contraception methods
* Those with occupations requiring use and/or operation of hazardous heavy equipment or professional drivers
* Patients for whom the potential risk outweighs the potential benefit in the opinion of the treating psychiatrist

Ages: 44 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-06-24 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles J Foulks, M.D., Study Chair — Central Texas Veterans Health Care System, Temple, TX
Locations (2):
- United States (2):
  - Central Texas Veterans Health Care System, Temple, TX, Temple, Texas
  - Central Texas Veterans Health Care System Waco VA Medical Center, Waco, TX, Waco, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment was very difficult.
Groups:
- Group 1: 60 mg of duloxetine in the AM for 20 weeks
  Duloxetine: serotonin norepinephrine reuptake inhibitor
  Placebo: Placebo
- Group 2: 300 mg of pregabalin in the PM for 20 weeks
  Pregabalin: alpha-2-alpha subunit calcium channel ligand
  Placebo: Placebo
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 0 (Unclear due to assignment records.) | 0 (Unclear due to assignment records.) | 0 (Unclear due to assignment records.)
Completed | 0 (The data on completion subjects is corrupted and not reliable for interpretation.) | 0 (The data on completion subjects is corrupted and not reliable for interpretation.) | 0 (The data on completion subjects is corrupted and not reliable for interpretation.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data collection was inaccurate and data are considered unreliable for evaluation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]
Pain

OUTCOME MEASURES:

1. Primary Outcome: Pain by Likert Scale
Description: Likert scale of pain rating
Time Frame: 120 days
Population: Data collection was inaccurate and data are considered unreliable for evaluation.
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Side Effects
Description: Side effects checklist
Time Frame: Assessed every 2 weeks
Population: Data collection was inaccurate and data are considered unreliable for evaluation.
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

3. Other Pre Specified Outcome: Multiple and Unreliable
Description: Reliability of measurement is highly suspect and data are not suitable for analysis.
Time Frame: Assessed every 2 weeks up to 34 weeks
Population: Data were inaccurately collected and are considered unreliable for interpretation.
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Entire study data are unreliable.
Description: Event collection appears to be inadequate and data are considered to be unreliable.
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was closed by the sponsor. Recruiting was very difficult and there were multiple irregularities in enrollment, data collection, and study management. The data are unreliable for interpretation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT01846182/Prot_SAP_000.pdf